CLINICAL TRIAL: NCT02123121
Title: Phase IIa Study of Resveratrol to Enhance Mitochondrial and Physical Function in Older Adults
Brief Title: Resveratrol to Enhance Vitality and Vigor in Elders
Acronym: REVIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB201400439 -A -N; 1R01AT007564-01 (NIH)
Record Dates: First submitted 2014-04-21; First posted 2014-04-25 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Mitochondrial Function; Physical Function
Keywords: Aging; Biogenesis; Cell Respiration; Elderly; Enzymes; Mitochondria; Mitochondrial DNA; Muscle Fatigue; Physical Function; Resveratrol
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vegetable cellulose (Placebo Comparator): Participants will orally consume one capsule of vegetable cellulose following each of their main meals (i.e. breakfast, lunch, and dinner) for 90 days.
  Interventions: Other: Vegetable cellulose; Other: All groups
- Resveratrol 1000 mg/day (Active Comparator): Participants will orally consume one capsule of Resveratrol following each of their main meals (i.e. breakfast, lunch, and dinner) totaling 1000 mg/day for 90 days.
  Interventions: Drug: Resveratrol 1000 mg/day; Other: All groups
- Resveratrol 1500 mg/day (Active Comparator): Participants will orally consume one capsule of Resveratrol following each of their main meals (i.e. breakfast, lunch, and dinner) totaling 1500 mg/day for 90 days.
  Interventions: Drug: Resveratrol 1500 mg/day; Other: All groups

INTERVENTIONS:
Drug: Resveratrol 1000 mg/day — Orally consume resveratrol 1000 mg/day capsule following each main meal (i.e. breakfast, lunch, and dinner), (i.e. take 3 capsules per day) for 90 Days.
  Arms: Resveratrol 1000 mg/day
Drug: Resveratrol 1500 mg/day — Orally consume resveratrol 1500 mg/day capsule following each main meal (i.e. breakfast, lunch, and dinner), (i.e. take 3 capsules per day) for 90 Days.
  Arms: Resveratrol 1500 mg/day
Other: Vegetable cellulose — Orally consume placebo vegetable cellulose capsule a day following each main meal (i.e. breakfast, lunch, and dinner), (i.e. take 3 capsules per day) for 90 Days.
  Other Names: Placebo
  Arms: Vegetable cellulose
Other: All groups — All Participants will have the following done: Physical Exams, Physical Measurements, Medical History, Questionnaires, Blood Samples, Tests of physical performance, and muscle tissue samples.

SUMMARY:
Resveratrol, a compound found in red wine and dark-skinned grapes, will improve the function of mitochondria (energy producing components) within the leg muscles of moderate functioning older adults.

The investigators will look at the role Resveratrol plays in improving physical function by studying the connection of changes in mitochondrial function and changes in physical function.

DETAILED DESCRIPTION:
An initial telephone screening indicated that the subject may be eligible to participate in the study. The first study visit ("Screening visit") will further determine if the subject is eligible to participate. Should the subject be eligible to participate in the study, the subject will be asked to participate in a daily resveratrol or placebo supplementation program for approximately 90 days. The subject will also be asked to return to the clinic for two additional assessment visits to monitor his/her safety and measure study results.

Details regarding the tests to be conducted during this screening visit and other study visits are described below. Visits will take place at the University of Florida Institute on Aging (IOA).

The Screening Visit is approximately 1.5 to 2 hours and will include:

1. Blood Draw: The subject is asked to fast before the appointment because blood will be collected during this visit. The investigator will collect approximately 2 tablespoons of blood. The purpose of this blood draw is to determine levels of certain compounds in the subject's blood that will help determine eligibility.
2. Questionnaires: The subject will be asked questions about medical history and medications as well as mood and will also be asked to complete a short test of memory and reasoning.
3. Physical Measurements: measurements of the subject's height, body weight, waist circumference, pulse, and blood pressure.
4. Physical Exam: A licensed health care provider will perform a brief physical exam to determine if it is safe to continue with the study. This exam will include a review of medical history, medications, and measurement of height, blood pressure, radial pulse, weight, and waist circumference.
5. Tests of physical performance: The subject will be asked to complete tests of physical ability that include:

   1. Walking at the usual pace for a distance of 13 feet (4 meters) two (2) separate times
   2. The subject will be asked to go from a standing to a sitting position, without using their arms. If the subject is able to perform this task, then they will be asked to stand up from and sit down on chair five (5) times as fast as possible.
   3. Maintaining balance while standing in three (3) different positions

Baseline Visit 1: Should the subject be eligible for the study, they will be asked to return to the clinic for the first baseline study visit. This visit is expected to take 2 to 3 hours and will include:

1. Measurement of pulse and blood pressure
2. Measurement of body weight and waist circumference
3. Collection of fasting blood samples
4. Questions about the subject's health
5. Tests of physical performance, including:

   1. Walking as fast and far as the subject can for 6 minutes
   2. Walking at subject's usual pace for a distance of 13 feet (4 meters) two (2) separate times
   3. Standing from a sitting position, without using their arms. If the subject is able to perform this task, then they will be asked to stand up from and sit down on chair five (5) times as fast as possible.
   4. Maintaining balance while standing in three (3) different positions.
   5. Assessment of lower-body muscle strength and endurance
6. Physical Activity Monitor: The subject will also be asked to wear an armband physical activity monitor during a typical seven day period to assess baseline physical activity habits. The monitor will be returned at Baseline Visit 2.

Baseline Visit 2 will take approximately 2 hours and will include:

1. Measurement of pulse and blood pressure before procedure
2. Muscle Tissue Sample: The procedure to collect muscle samples will be performed by a licensed healthcare provider with experience conducting the procedure. The procedure includes numbing a small area on the thigh with a local anesthetic and then using a needle about the size of a pen to collect a small amount of muscle tissue approximately equal to the size of the head of a pencil eraser.

   After the tissue sample is taken, the subject will receive detailed instruction on how to care for the incision site. Several follow-up phone assessments will be made inquiring about any problems that the subject may be experiencing related to the procedure.
3. Measurement of pulse and blood pressure after procedure
4. Randomization: Subjects who are eligible and safe to continue with the study, will be randomly assigned to one of three conditions: (1) resveratrol (1000 mg/day) (2) resveratrol (1500 mg/day) or (3) placebo (vegetable cellulose).
5. The subject will be provided with a supply of the study drug capsules of at least 30 days and will be asked to return any remaining study drug capsules to the clinic at the next appointment. Subjects will be asked to orally consume one study drug capsule following each main meal (i.e. breakfast, lunch and dinner) with a glass of water.

30-Day & 60-Day Visits last approximately 1 hour and include:

1. Collection of fasting blood samples
2. Measurement of pulse and blood pressure
3. Measurement of weight and waist circumference
4. Update medical history and ask questions about any adverse experiences the subject may have had since the last visit
5. Counting of any remaining study drug capsules that were not taken since last visit
6. Providing the subject with study drug capsules needed until the next study visit

90-Day Visit 1 is similar to the Baseline 1 visit and will last approximately 2-3 hours. This visit includes:

1. Measurement of pulse and blood pressure
2. Measurement of body weight and waist circumference
3. Collection of fasting blood samples
4. Update medical history and ask questions about any adverse experiences the subject may have had since last visit
5. Counting of any remaining study drug capsules that were not taken since last visit
6. Tests of physical performance, including:

   1. Walking as fast and far as possible for 6 minutes
   2. Walking at usual pace for a distance of 13 feet (4 meters) two (2) separate times
   3. Standing from a sitting position, without using arms. If the subject is able to perform this task, he/she will be to stand up from and sit down on chair five (5) times as fast as possible.
   4. Maintaining balance while standing in three (3) different positions.
   5. Assessment of lower-body muscle strength and endurance
7. The subject will receive an armband physical activity monitor to wear for seven days, and will be asked to return this monitor at the 90-Day Visit 2.

90-Day Visit 2 will be similar to the Baseline 2 visit and will last approximately 1.5 to 2 hours.

1. Procedure to collect muscle tissue sample (as described in Baseline 2)
2. Counting of any remaining study drug capsules that were not taken since last visit.

Follow-Up 10-Day & 30-Day Visits are approximately 30 minutes to 1 hour

1. Measurement of pulse and blood pressure
2. Collection of fasting blood samples
3. Update medical history and ask questions about any adverse experiences the subject may have had since last visit

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand study procedures and to comply with them for the entire length of the study;
* Age 65 years and older;
* Moderate to high functioning (i.e. a summary score of 4 - 10 on the Short Physical Performance Battery [SPPB]);
* Body Mass Index (BMI) range: 20-39.9 kg/m2;
* Willingness to undergo all testing procedures.

Exclusion Criteria:

* Failure to provide informed consent;
* Allergy/sensitivity to grapes or Japanese knotweed;
* Current dietary supplementation of grape seed extract or ginko biloba;
* Consumption of ≥ 8 oz. of red wine/dealcoholized red wine/red or purple grape juice more than once weekly;
* Consumption of any dietary supplements containing resveratrol, quercetin, or P. cuspidatum in the previous 90 days;
* Active treatment for cancer, stroke (< 6 months), peripheral vascular disease, coronary artery disease, myocardial infarction (< 6 months), congestive heart failure (stage III or IV), valvular heart disease, major psychiatric disease, severe anemia (blood levels of Hemoglobin < 8 g/dl), liver or renal disease, diabetes, severe osteoarthritis, blindness or deafness, fracture in upper or lower extremity ( < 6 months), upper or lower extremity amputation, or Parkinson's disease;
* Cognitive impairment (i.e. Mini Mental Status Exam ≤ 23);
* History of significant head injury;
* Physical activity (i.e. running, bicycling, etc.) ≥ 120 min/week;
* Excessive alcohol use (> 2 drinks/day) or alcohol abuse (> 5 drinks/day for males, or > 4 drinks/day for females);
* History of substance abuse within the past six months;
* Mood disorder (i.e. Center for Epidemiological Studies - Depression (CES-D) ≥ 16);
* History of tobacco use within the past three years;
* Resting heart rate > 120 bpm at screening visit;
* Systolic blood pressure > 160 mm Hg at screening visit;
* Diastolic blood pressure > 90 mm Hg at screening visit;
* Fasting glucose ≥ 126 mg/dL at screening visit;
* Abnormalities in blood chemistry parameters, defined by blood chemistry marker outside of healthy range);
* Current use of anabolic treatments (e.g. growth hormone or testosterone), anticholinesterase inhibitor (e.g. Aricept), hormone replacement (e.g. Estrogen), or anticoagulant therapies (note: aspirin use (≤ 81mg/day) is permitted);
* Participation in another clinical trial, or has received an investigational product within 30 days prior to screening/enrollment;
* Refuse to refrain from CoQ10 or alpha-lipoic acid while enrolled in the study.

Temporary Exclusion Criteria

* Recent bacterial/viral infection (< 2 weeks);
* Acute febrile illness in past 2 months;
* High blood pressure (i.e. ≥ 140/90 mm Hg but ≤ 160/90) at the screening visit;
* Major surgery or hip/knee replacement (< 6 months).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Anton, Ph.D., Principal Investigator — University of Florida
Locations (1):
- UF Institute on Aging Clinical and Translational Research Building, Gainesville, Florida, United States

REFERENCES:
- See also: University of Florida Institute on Aging — http://aging.ufl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Started | 20 | 21 | 19
Completed | 18 | 20 | 16
Not Completed | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day | Total
Number analyzed (Participants) | 20 | 21 | 19 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.72 (5.94) | 73.4 (5.63) | 73.18 (5.78) | 74.1 (5.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 13 | 37
  Male | 8 | 9 | 6 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 16 | 18 | 13 | 47
  Non-Hispanic Black | 1 | 3 | 6 | 10
  Non-Hispanic Other | 1 | 0 | 0 | 1
  Hispanic | 2 | 0 | 0 | 2
Marital Status [Count of Participants; unit: Participants]
  Never Married | 1 | 0 | 1 | 2
  Married | 10 | 11 | 5 | 26
  Separated/Divorced/Widowed | 8 | 10 | 13 | 31
  Other | 1 | 0 | 0 | 1
Live Alone [Count of Participants; unit: Participants]
  Yes | 6 | 5 | 7 | 18
  No | 14 | 16 | 12 | 42
Highest Level of Education [Count of Participants; unit: Participants]
  High School/Equivalent | 5 | 4 | 5 | 14
  College | 5 | 9 | 9 | 23
  Post-Graduate | 7 | 8 | 5 | 20
  Other | 3 | 0 | 0 | 3
Income [Count of Participants; unit: Participants]
  <$35,000 | 9 | 9 | 7 | 25
  $35,000-$74,999 | 7 | 8 | 9 | 24
  >=$75,000 | 3 | 2 | 2 | 7
  Don't Know/Refused | 1 | 2 | 1 | 4
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (4.4) | 27.8 (3.8) | 29.3 (5.3) | 28.4 (4.5)
Physical Activity [Mean (Standard Deviation); unit: minutes in moderate/vigorous activity] — Population: Dropout occurred.
  minutes in moderate/vigorous activity
    number analyzed (Participants) | 17 | 20 | 18 | 55
    (all) | 44.0 (26.5) | 44.2 (22.5) | 49.2 (22.5) | 45.8 (23.8)
Six Minute Walk [Mean (Standard Deviation); unit: meters per second] — Test, where participants will be asked to walk as far and fast as possible for 6-min on a 40 m track
  meters per second | 1.2 (0.3) | 1.2 (0.2) | 1.1 (0.1) | 1.2 (0.2)
Short Physical Performance Battery (SPPB) [Mean (Standard Deviation); unit: units on a scale (0-12)] — The SPPB is designed to assess lower-extremity function by measuring three timed subtests: five timed repetitive chair stands, standing balance (i.e. hold tandem and semi-tandem foot position for 10 seconds), and gait speed during a 4 m walk at one's usual pace. Each subtest is scored from 0 to 4, with 0 indicating inability to complete test, and 4 indicating maximal performance. A summary score from 0 to 12 is calculated for the SPPB, where higher scores indicate better physical function.
  units on a scale (0-12) | 10.6 (2.0) | 11.0 (1.5) | 11.3 (0.7) | 11.0 (1.4)
Knee Flexion [Mean (Standard Deviation); unit: Peak Torque (nm)] — This test involves using an isokinetic dynamometer set at 90 degrees per second. Participants will perform 50 maximal knee extension and flexion concentric repetitions, which will be administered by trained and certified research assistants.
  Peak Torque (nm) | 32.2 (14.0) | 37.4 (15.8) | 31.2 (12.4) | 33.6 (13.7)
Waist Circumference [Mean (Standard Deviation); unit: Centimeters] | 98.4 (9.3) | 99.2 (10.8) | 100.1 (18.4) | 99.2 (12.8)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 98.6 (9.5) | 92.4 (7.4) | 94.3 (9.1) | 95.1 (8.7)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74.7 (9.3) | 77.0 (8.6) | 75.4 (7.9) | 75.4 (8.6)
PGC-1 alpha [Mean (Standard Deviation); unit: arbitrary units] — Peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α) is a protein that in humans is encoded by the PPARGC1A gene.
  arbitrary units | 0.48 (0.12) | 0.52 (0.16) | 0.55 (0.19) | 0.52 (0.16)
SIRT-1 [Mean (Standard Deviation); unit: arbitrary units] | 0.7 (0.25) | 0.79 (0.29) | 0.71 (0.18) | 0.73 (0.24)
SIRT-3 [Mean (Standard Deviation); unit: arbitrary units] | 0.37 (0.14) | 0.42 (0.14) | 0.43 (0.18) | 0.41 (0.15)
Mitochondrial DNA Content [Mean (Standard Deviation); unit: ratio] — Mitochondrial DNA content is measured based on the ratio of the mitochondrial genome to nuclear genome ratio (Mt/N)
  ratio | 384.3 (139.9) | 409.1 (127.4) | 329.3 (86.1) | 374.2 (117.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mitochondrial Respiration in Muscle
Description: Change in mitochondrial respiration (State 3) in muscle samples of moderate-to-low functioning older adults from baseline to post-test (90 days).
Time Frame: Baseline to 90 Days
Measure: Mean (95% Confidence Interval); unit: nmol O2/s/mg wwt
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
nmol O2/s/mg wwt | -3.05 [-9.90 to 3.81] | -4.82 [-11.03 to 1.38] | -4.56 [-12.07 to 2.94]

2. Primary Outcome: Change From Baseline in Cytochrome Oxidase (COX) in Muscle Samples
Description: Change in cytochrome oxidase (COX) in muscle samples of moderate-to-low functioning in older adults from baseline to post-test (90 days).
Time Frame: Baseline to 90 days
Population: Population measured after participant dropout.
Measure: Mean (Standard Deviation); unit: nmol/min/mg/protein
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 13 | 17 | 11
nmol/min/mg/protein | 109.4 (58.26) | 126.7 (34.10) | 121.2 (48.46)

3. Primary Outcome: Change From Baseline in Citrate Synthase (CS) Enzymes in Muscle Samples
Description: Change in citrate synthase (CS) enzymes in muscle samples of moderate-to-low functioning in older adults from baseline to post-test (90 days).
Time Frame: Baseline to 90 Days
Measure: Mean (95% Confidence Interval); unit: nmol/min/mg protein
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
nmol/min/mg protein | -0.02 [-0.25 to 0.20] | 0.08 [-0.13 to 0.29] | -0.09 [-0.34 to 0.16]

4. Primary Outcome: Change From Baseline in Mitochondrial DNA Content in Muscle Samples
Description: Change in mitochondrial DNA content in muscle samples of moderate-to-low functioning in older adults from baseline to post-test (90 days).
Time Frame: Baseline and 90 Days
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
Ratio | 2.71 [-43.58 to 49.01] | 7.13 [-36.80 to 51.06] | -7.31 [-58.32 to 43.71]

5. Secondary Outcome: Change From Baseline in PGC-1α Muscle Protein Levels
Description: Change in muscle protein levels, such as PGC-1α (primary outcome) in muscle samples of moderate-to-low functioning older adults from baseline to post-test (90 days). Arbitrary units are used for measurement as it is common for protein expression data since we do not measure absolute content of a specific protein within a sample.
Time Frame: Baseline to 90 Days
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
arbitrary units | -0.10 [-0.15 to -0.04] | -0.12 [-0.17 to -0.07] | -0.07 [-0.13 to -0.01]

6. Secondary Outcome: Change From Baseline in Walking Speed.
Description: Change in physical function, such as walking speed from baseline to post-test (90 days). The Six Minute Walk Test was used to measure data and involved participants being asked to walk as far and as fast as possible for 6-minutes on a 40m track.
Time Frame: Baseline to 90 Days
Measure: Mean (95% Confidence Interval); unit: m/s
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
m/s | 0.03 [0.01 to 0.08] | 0.06 [0.01 to 0.10] | 0.04 [0.00 to 0.09]

7. Secondary Outcome: Blood Glucose Level
Description: Change in levels of blood glucose (metabolic risk factor) from baseline to post-test (90 days).
Time Frame: Baseline to 90 Days
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
mg/dL | 9.49 [2.3 to 16.67] | 0.74 [-2.02 to 3.49] | 2.94 [-2.64 to 8.51]

8. Secondary Outcome: Physical Activity Levels
Description: Change in levels of spontaneous physical activity from baseline to post-test (90 days). Measured using an accelerometer which is a wearable device that captures acceleration (counts) in real time, in multiple planes. Can be used to measure energy expenditure or stationary activity levels.
Time Frame: Baseline to 90 Days
Measure: Mean (Standard Deviation); unit: Counts per minute
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
Counts per minute | 167.0 (99.6) | 153.1 (69.2) | 170.9 (62.9)

9. Secondary Outcome: Change From Baseline in AMPK Muscle Protein Levels.
Description: Change in muscle protein levels, such as AMPK in muscle samples of moderate-to-low functioning older adults from baseline to post-test (90 days). Arbitrary units are used for measurement as it is common for protein expression data since we do not measure absolute content of a specific protein within a sample.
Time Frame: Baseline to 90 Days
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 13 | 13 | 11
arbitrary units | 0.42 (0.37) | 0.72 (0.43) | 1.50 (2.44)

10. Secondary Outcome: Change From Baseline in Sirtuins (SIRT1) Muscle Protein Levels.
Description: Change in muscle protein levels, such as sirtuins (SIRT1), in muscle samples of moderate-to-low functioning older adults from baseline to post-test (90 days). Arbitrary units are used for measurement as it is common for protein expression data since we do not measure absolute content of a specific protein within a sample.
Time Frame: Baseline to 90 Days
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
arbitrary units | 0.03 [-0.04 to 0.10] | 0.00 [-0.06 to 0.07] | 0.01 [-0.06 to 0.08]

11. Secondary Outcome: Change From Baseline in Physical Performance
Description: Change in Short Physical Performance Battery (SPPB) Test Total Score on a scale of 0-12 from baseline to post-test (90 days). Lower scores indicate more mobility limitations while higher scores indicate minimal to no mobility limitations.
Time Frame: Baseline to 90 Days
Measure: Mean (95% Confidence Interval); unit: units on a scale 0-12
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
units on a scale 0-12 | 0.18 [-0.13 to 0.50] | -0.08 [-0.39 to 0.22] | 0.06 [-0.27 to 0.38]

12. Secondary Outcome: Change From Baseline in Sirtuins (SIRT3) Muscle Protein Levels.
Description: Change in muscle protein levels, such as sirtuins (SIRT3), in muscle samples of moderate-to-low functioning older adults from baseline to post-test (90 days). Arbitrary units are used for measurement as it is common for protein expression data since we do not measure absolute content of a specific protein within a sample.
Time Frame: Baseline to 90 days
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
Number analyzed (Participants) | 20 | 21 | 19
arbitrary units | 0.01 [-0.02 to 0.04] | 0.01 [-0.02 to 0.04] | -0.01 [-0.04 to 0.02]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Vegetable Cellulose | Resveratrol 1000 mg/Day | Resveratrol 1500 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 14/20 | 12/21 | 16/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vegetable Cellulose (N=20) | Resveratrol 1000 mg/Day (N=21) | Resveratrol 1500 mg/Day (N=19)
Diarrhea, Burning in Stomach, Loose Stool, Nausea and Vomiting, Constipation, (Gastrointestinal disorders) | 5 | 9 | 11
General Issues (General disorders) | 10 | 2 | 10 — Patients experiencing adverse events including: low energy, headaches, seasonal allergies
Muscle soreness, joint inflammation and pain, hand surgery (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4
Bronchitis, conjunctivitis, common cold, bacterial and fungal infections (Infections and infestations) | 9 | 1 | 9
Increased urination urge, UTI, and kidney stones (Renal and urinary disorders) | 1 | 3 | 1
Abnormal liver function values (Hepatobiliary disorders) | 0 | 0 | 1
Tinnitis in ear (Ear and labyrinth disorders) | 0 | 0 | 1
Significantly low platelet and white blood cell count (Blood and lymphatic system disorders) | 0 | 0 | 1
Product issue (General disorders) | 0 | 1 | 0 — Patient reported feeling a "fullness" in his throat after swallowing pills
Atrial Fibrillation and irregular heart beat (Cardiac disorders) | 2 | 0 | 0
Snake Bite (Social circumstances) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT02123121/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02123121/ICF_001.pdf